CLINICAL TRIAL: NCT06761313
Title: Triplenex (triple Fixed Combination) Use Evaluation in Patients with Glaucoma: Randomized Clinical Trial
Brief Title: Triplenex (triple Fixed Combination) Use Evaluation in Patients with Glaucoma
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Lilian França Machado, Medical Doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.261.282
Record Dates: First submitted 2024-12-13; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma; Quality of Life (QOL)
Keywords: Glaucoma; Triplenex; Triple combination; QoL; Addherence
MeSH Terms: conditions — Glaucoma | interventions — Timolol; Bimatoprost

STUDY DESIGN:
Intervention Model Description: In this clinical trial approved by the Unifesp Etical and Research Comitte, volunteer glaucoma patients will be recruited from Unifesp Glaucoma Sector and VerMais Glaucoma Sector. They will be randomly divided em two groups,Group I is going to be treated with Triplenex (1 drop twice a day) and Grupo II with Brimonidine Tartarate (1 drop twice a day), Timolol Maleate (1 drop twice a day) and Bimatoprost (1 drop at night). At baseline visit a complete ophthalmolgical exam will be performed along with three questionnaires ("Ocular Surface Disease Index", "Glaucoma Treatment Compliance Assessment Tool" and "National Eye Institute Visual Function Questionnaire"),retinography, visual field, optic nerve OCT in all patients. This procedure will be repeated at baseline and within 4, 8, 12 weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I: Triplenex (Triple Fixed Combination Eyedrop) (Experimental): After the visit during which their previous hypotensive eye drops are suspended, thus determining the baseline intraocular pressure and the ocular surface at this moment, the patients will be randomized. The experimental group (Group I) is going to be treated with Triplenex (a combination of the three drugs included in the control group), patients will be instructed to use 1 drop twice a day .
  Interventions: Drug: Triple combination formula
- Group II: Brimonidine Tartarate 0.2%, Timolol Maleate 0.5%, Bimatoprost 0.03% (Other): After the visit during which their previous hypotensive eye drops are suspended, thus determining the baseline intraocular pressure and the ocular surface at this moment, the patients will be randomized. The control group (Group II) is going to be treated with a combination of three separated eyedrops: Brimonidine Tartarate 0.2%,Timolol Maleate 0.5%, Bimatoprost 0.03%. The dosage for the eye drops Brimonidine Tartarate and Timolol Maleate will be twice a day. The drug Bimatoprost is advised to be instilled once at night. The use of the combination of the three separate drugs is instructed with a time interval of at least 10 minutes between each class of eye drop.
  Interventions: Drug: Bimatoprost .03% sterile ophthalmic solution

INTERVENTIONS:
Drug: Triple combination formula — Individuals will be randomly divided em two groups,Group I is going to be treated with Triplenex (1 drop twice a day) and Grupo II with Brimonidine Tartarate (1 drop twice a day), Timolol Maleate (1 drop twice a day) and Bimatoprost (1 drop at night). At baseline visit a complete ophthalmolgical exam will be performed along with three questionnaires ("Ocular Surface Disease Index", "Glaucoma Treatment Compliance Assessment Tool" and "National Eye Institute Visual Function Questionnaire"),retinography, visual field, optic nerve OCT in all patients. This procedure will be repeated at baseline and within 4, 8, 12 weeks.
  Other Names: Maleate Timolol 0.5%, Brimonidine Tartarate 0.2%, Bimatoprost 0.03%
  Arms: Group I: Triplenex (Triple Fixed Combination Eyedrop)
Drug: Bimatoprost .03% sterile ophthalmic solution — Individuals will be randomly divided em two groups,Group I is going to be treated with Triplenex (1 drop twice a day) and Grupo II with Brimonidine Tartarate 0.2%(1 drop twice a day), Timolol Maleate 0.5% (1 drop twice a day) and Bimatoprost 0.3% (1 drop at night). At the first visit a complete ophthalmolgical exam which includes ocular surface items (conjunctival hiperemia, keratitis and tear film break up time). Questionnaires are performed ("Ocular Surface Disease Index", "Glaucoma Treatment Compliance Assessment Tool" and "National Eye Institute Visual Function Questionnaire") to assess information about ocular surface adverse effects, quality of life and treatment adherence. Glaucoma exams as retinography, perimetry, optic nerve OCT (optical coherence tomography), central corneal thickness are performed on all patients to evaluate disease's control. This procedure will be repeated at all visits: baseline and within 4, 8, 12 weeks.
  Other Names: Timolol Maleate 0.5%; Brimonidine Tartarate 0.2%; Bimatoprost 0.03%
  Arms: Group II: Brimonidine Tartarate 0.2%, Timolol Maleate 0.5%, Bimatoprost 0.03%

SUMMARY:
This project purpose is to evaluate the effectiveness, ocular surface quality, medication adherence and quality of life in 46 glaucoma patients in use of three separate drugs (Bimatoprost 0.3%, Timolol Maleate 0.5% and Brimonidine Tartrate 0.2%) comparing with triple combination, Triplenex. In this clinical trial approved by the Unifesp Etical and Research Comitte, volunteer glaucoma patients will be recruited from Unifesp Glaucoma Sector and VerMais Glaucoma Sector. They will be randomly divided em two groups,Group I is going to be treated with Triplenex (1 drop twice a day) and Grupo II with Brimonidine Tartarate (1 drop twice a day), Timolol Maleate (1 drop twice a day) and Bimatoprost (1 drop at night). At baseline visit a complete ophthalmolgical exam will be performed along with three questionnaires ("Ocular Surface Disease Index", "Glaucoma Treatment Compliance Assessment Tool" and "National Eye Institute Visual Function Questionnaire"),retinography, visual field, optic nerve OCT in all patients. This procedure will be repeated at baseline and within 4, 8, 12 weeks.

DETAILED DESCRIPTION:
This clinical study aims to compare the use of the hypotensive eye drop Triplenex, a fixed triple combination (currently available only in Brazil, Mexico, and Chile), with the globally recognized combination of the same drugs administered separately. The combination of the eye drops Bimatoprost 0.3%, Timolol Maleate 0.5%, and Brimonidine Tartrate 0.2% in separate vials is traditionally used in patients with difficult intraocular pressure control or advanced glaucoma that requires a low target pressure for proper disease management. The fixed triple combination intends to improve patient adherence while maintaining the efficacy of intraocular pressure control and progression of glaucoma. This study arises in the context of a lack of literature comparing Triplenex to the three original drugs and the absence of data on its influence on adherence, ocular surface, and the quality of life in the daily lives of glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosed glaucoma
* above 18 years old
* in use of at least 3 different glaucoma eyedrops classes
* informed consent form granted

Exclusion Criteria:

* secundary glaucoma
* previous ocular surface disease
* previous intraocular surgeries (except cataract)
* previous ocular trauma
* current use of contact lenses use
* current use of steroids or systemic medications that may change ocular surface
* any study's drug intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-02-26 (Estimated)

PRIMARY OUTCOMES:
Triplenex (triple fixed combination) use evaluation in patients with Glaucoma: randomized clinical trial | From enrollment to the end of treatment at 6 months
  Compare the efficacy of Triplenex (fixed triple combination) to the same substances separated into three eye drops (Bimatoprost 0.03%, Timolol Maleate 0.5%, and Brimonidine Tartrate 0.2%). The comparison of efficacy between the groups will be evaluated based on the reduction of intraocular pressure and control of glaucoma progression.
Triplenex (triple fixed combination) use evaluation in patients with Glaucoma: randomized clinical trial | From enrollment to the end of treatment at 6 months
  Compare the adverse effects of Triplenex (fixed triple combination) to the same substances separated into three eye drops (Bimatoprost 0.03%, Timolol Maleate 0.5%, and Brimonidine Tartrate 0.2%). The side effects will be mesured by the following assessments: ocular surface assessment (conjunctival hyperemia, tear film break-up time, keratitis) and (Ocular Surface Disease Index) questionnaire. Conjunctival hyperemia and keratitis are measured on a 5-level scale, with the last level being the worst classification. Tear film break-up time is measured in time from 0 to 10 seconds, the longer the tear film takes to break the better the result.

SECONDARY OUTCOMES:
Triplenex (triple fixed combination) use evaluation in patients with Glaucoma: randomized clinical trial | From enrollment to the end of treatment at 6 months
  Compare the adherence to the treatment of glaucoma patients using the fixed combination to the use of the same three drugs separately. A compliance questionnaire (Glaucoma Treatment Compliance Assessment Tool) score will be used in comparison between groups.
Triplenex (triple fixed combination) use evaluation in patients with Glaucoma: randomized clinical trial | From enrollment to the end of treatment at 6 months
  Compare the quality of life of patients using the triple fixed combination to the use of the same three drugs separately. A quality of life questionnaire (Visual Function Questionnaire-25) will be performed every visit generating a score that will be used in the comparison between groups, in this scale a higher score means better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Gracitelli, Affiliate Professsor, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data sheet that does not identify the patient, and also the statistic analyses.

REFERENCES:
- [Background] The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):75-92. doi: 10.1016/s1542-0124(12)70081-2. PMID 17508116
- [Background] Goldberg I, Clement CI, Chiang TH, Walt JG, Lee LJ, Graham S, Healey PR. Assessing quality of life in patients with glaucoma using the Glaucoma Quality of Life-15 (GQL-15) questionnaire. J Glaucoma. 2009 Jan;18(1):6-12. doi: 10.1097/IJG.0b013e3181752c83. PMID 19142128
- [Background] Baffa Ldo P, Ricardo JR, Dias AC, Modulo CM, Braz AM, Paula JS, Rodrigues Mde L, Rocha EM. Tear film and ocular surface alterations in chronic users of antiglaucoma medications. Arq Bras Oftalmol. 2008 Jan-Feb;71(1):18-21. doi: 10.1590/s0004-27492008000100004. PMID 18408831
- [Background] Skalicky SE, Goldberg I, McCluskey P. Ocular surface disease and quality of life in patients with glaucoma. Am J Ophthalmol. 2012 Jan;153(1):1-9.e2. doi: 10.1016/j.ajo.2011.05.033. Epub 2011 Aug 26. PMID 21872203
- [Background] Fechtner RD, Godfrey DG, Budenz D, Stewart JA, Stewart WC, Jasek MC. Prevalence of ocular surface complaints in patients with glaucoma using topical intraocular pressure-lowering medications. Cornea. 2010 Jun;29(6):618-21. doi: 10.1097/ICO.0b013e3181c325b2. PMID 20386433
- [Background] Mangione CM, Lee PP, Gutierrez PR, Spritzer K, Berry S, Hays RD; National Eye Institute Visual Function Questionnaire Field Test Investigators. Development of the 25-item National Eye Institute Visual Function Questionnaire. Arch Ophthalmol. 2001 Jul;119(7):1050-8. doi: 10.1001/archopht.119.7.1050. PMID 11448327
- [Background] Newman-Casey PA, Robin AL, Blachley T, Farris K, Heisler M, Resnicow K, Lee PP. The Most Common Barriers to Glaucoma Medication Adherence: A Cross-Sectional Survey. Ophthalmology. 2015 Jul;122(7):1308-16. doi: 10.1016/j.ophtha.2015.03.026. Epub 2015 Apr 24. PMID 25912144
- [Background] Olthoff CM, Schouten JS, van de Borne BW, Webers CA. Noncompliance with ocular hypotensive treatment in patients with glaucoma or ocular hypertension an evidence-based review. Ophthalmology. 2005 Jun;112(6):953-61. doi: 10.1016/j.ophtha.2004.12.035. PMID 15885795
- [Background] Mansberger SL, Sheppler CR, McClure TM, Vanalstine CL, Swanson IL, Stoumbos Z, Lambert WE. Psychometrics of a new questionnaire to assess glaucoma adherence: the Glaucoma Treatment Compliance Assessment Tool (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2013 Sep;111:1-16. PMID 24072942
- [Background] Belfort R Jr, Paula JS, Lopes Silva MJ, Della Paolera M, Kim T, Chen MY, Goodkin ML. Fixed-combination Bimatoprost/Brimonidine/Timolol in Glaucoma: A Randomized, Masked, Controlled, Phase III Study Conducted in Brazil☆. Clin Ther. 2020 Feb;42(2):263-275. doi: 10.1016/j.clinthera.2019.12.008. Epub 2020 Feb 20. PMID 32089329
- [Background] Hartleben C, Parra JC, Batoosingh A, Bernstein P, Goodkin M. A Masked, Randomized, Phase 3 Comparison of Triple Fixed-Combination Bimatoprost/Brimonidine/Timolol versus Fixed-Combination Brimonidine/Timolol for Lowering Intraocular Pressure. J Ophthalmol. 2017;2017:4586763. doi: 10.1155/2017/4586763. Epub 2017 Sep 19. PMID 29057117